CLINICAL TRIAL: NCT04159740
Title: Microbiome and Immunologic Analysis of the Lower and Upper Female Reproductive Tract in Women With Endometriosis
Brief Title: Microbiome and Immunologic Analysis - Women With Endometriosis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marina R. Walther-Antonio, Assistant Professor of Surgery, Mayo Clinic
Other Study IDs: 18-011885
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis - Cases: Premenopausal women with suspected endometriosis, planning to undergo laparoscopic surgery.
  Interventions: Other: Tissue and blood collection
- Controls: Premenopausal women without endometriosis, planning to undergo laparoscopic surgery for non-cancer indications including elective salpingectomy, tubal ligation or surgical procedures for abnormal uterine bleeding
  Interventions: Other: Tissue and blood collection

INTERVENTIONS:
Other: Tissue and blood collection — Tissue and swab (cells) collection for microbiome analysis. Blood collection for immune markers.

SUMMARY:
The primary goal of this study is to assess differences in the microbiome between women with and without endometriosis.

A second goal of this study is to assess immunologic differences between the eutopic (within the uterus) and ectopic (outside of the uterus) endometrial tissue in women with endometriosis.

In order to investigate these areas of interest, 25 women with endometriosis and 25 women without endometriosis will be enrolled. All women will be undergoing a previously scheduled surgical procedure at which time presence or absence of endometriosis will be confirmed and specimens will be obtained.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynecologic condition where implants of endometrial glands and stroma are present outside of the uterus. It occurs in 6-10% of women of reproductive age and is characterized by dysmenorrhea, chronic pelvic pain, dyspareunia, or infertility. In addition to symptom burden, there are significant direct costs related to diagnosis and treatment of disease, as well as indirect costs related to absenteeism from school and work, loss of productivity, and unemployment. The estimated national economic burden in the United States related to these costs is approximately 78 billion dollars per year. While clinical signs and symptoms may be suggestive of endometriosis, the gold standard for diagnosis requires surgical confirmation of disease.

The pathogenesis of endometriosis is complex and likely multifactorial with genetic, epigenetic, environmental, and immunologic factors. An increasing number of studies have also suggested the role of the microbiome in human health and development of disease. This study aims to investigate possible differences in the microbiome and immunologic factors that could contribute to pathogenesis of this disease. Findings from this study could potentially contribute to the development of of a less invasive, non-surgical diagnostic test for endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Females, age 18 years or older
* Undergoing laparoscopy (conventional or robotic) with or without hysterectomy for non-cancer indications and including women from two groups:
* Suspected endometriosis
* Elective salpingectomy or tubal ligation or abnormal uterine bleeding
* Understands study procedures
* Willing and able to provide signed informed consent

Exclusion Criteria:

* Postmenopausal
* Currently pregnant or lactating
* Prior hysterectomy or oophorectomy
* Undergoing hysterectomy via vaginal or abdominal approach
* Undergoing hysterectomy or laparoscopy for suspected malignancy
* Use of antibiotics within 2 weeks prior to surgery
* Use of hormone therapy for endometriosis or contraception within 4 weeks prior to surgery
* Diagnosis or treatment of vaginitis during the past 6 months prior to surgery
* Personal history of autoimmune or inflammatory disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women with or without endometriosis, planning to undergo laparoscopic surgery for non-cancer indications.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Microbiome composition in genital tract and gastrointestinal tract | At time of surgery

SECONDARY OUTCOMES:
Immunostaining of eutopic and ectopic endometrium for immune factors, immune cells, and fibrosis | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marina R Walther-Antonio, Ph.D., Principal Investigator — Mayo Clinic; Adela G Cope, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials